CLINICAL TRIAL: NCT06122649
Title: A Phase 3b, Multicenter, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Study of Apremilast 30 mg Twice Daily in Chinese Subjects With Moderate to Severe Plaque-type Psoriasis
Brief Title: A Study to Investigate Efficacy and Safety of Apremilast 30 mg Twice Daily (BID) in Chinese Participants With Moderate to Severe Plaque-type Psoriasis (PsO)
Acronym: ESSENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20200250
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
Keywords: Apremilast; Dermatology
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo-controlled Treatment Phas (Experimental): Participants are randomized in a 1:1 ratio to take either apremilast or placebo BID for 16 weeks.
  Interventions: Drug: apremilast; Drug: Placebo
- Active Treatment Phase (Experimental): Participants who received placebo during the placebo-controlled treatment phase will receive apremilast BID for 36 weeks. Participants who took apremilast will continue receiving it BID for 36 weeks.
  Interventions: Drug: apremilast

INTERVENTIONS:
Drug: apremilast — Oral tablet
  Other Names: Otezla®
Drug: Placebo — Oral tablet
  Arms: Placebo-controlled Treatment Phas

SUMMARY:
The study aims to evaluate the clinical efficacy of oral apremilast 30 mg BID compared with placebo in Chinese participants with moderate to severe PsO

ELIGIBILITY:
Inclusion Criteria

* Chinese participants aged ≥18.
* Diagnosis of chronic, stable moderate to severe plaque PsO for ≥ 12 months before screening. The participant must have sPGA score ≥ 3, PASI score ≥ 12, and BSA involvement ≥ 10% at both screening and baseline (week 0).
* Participant is a candidate for phototherapy and/or systemic therapy. Exclusion Criteria
* Psoriasis flare within 4 weeks of screening.
* Evidence of skin conditions that would interfere with evaluations of the effect of study medication on psoriasis.
* Prior medical history of suicide attempt at any time in the participant's lifetime before screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
* Participant has a malignancy or history of malignancy or myeloproliferative or lymphoproliferative disease within the past 3 years.
* Active tuberculosis or a history of incompletely treated tuberculosis.
* History of human immunodeficiency virus (HIV) infection.
* Prior treatment with apremilast.
* Female participants of childbearing potential unwilling to use protocol specified method of contraception.
* Female participants who are breastfeeding or who plan to breastfeed.
* Female participants planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants Achieving at least a 75% Reduction (Improvement) From Baseline in Psoriasis Area and Severity Index (PASI) at Week 16 | Week 16

SECONDARY OUTCOMES:
Number of Participants Achieving a Static Physician's Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) and with ≥ 2-point Reduction From Baseline at Week 16 | Baseline and Week 16
Number of Participants Achieving ≥ 4-point Reduction (Improvement) From Baseline in the Whole Body Itch Scale (NRS) Score at Week 16 | Baseline and Week 16
Number of Participants with Baseline Scalp Physician's Globa Assesment (ScPGA) of ≥ 2 Achieving a Clear (0) or Almost Clear (1) ScPGA and with ≥ 2-point Reduction From Baseline and at Week 16 | Baseline and Week 16
Percent Change of PASI From Baseline at Week 16 | Baseline and Week 16
Percent Change From Baseline in Affected Body Surface Area (BSA) at Week 16 | Baseline and Week 16
Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 16 | Baseline and Week 16
Number of Participants who Have a Baseline Scalp Itch NRS ≥ 4 and Achieving ≥ 4-point Reduction (Improvement) From Baseline in Scalp Itch NRS at Week 16 | Baseline and Week 16
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Baseline to Week 52
  TEAEs are any event that occurred after the participant received study treatment. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs.
Plasma Concentration of Apremilast | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (21):
- China (21):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang First Peoples Hospital, Nanyang, Henan
  - Yichang Central Peoples Hospital, Yichang, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Changshu No2 Peoples Hospital, Suzhou, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Provincial Hospital For Skin Diseases,Shandong First Medical University, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Peoples Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2 ) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com